CLINICAL TRIAL: NCT00423059
Title: Histologic Changes of Fibrovascular Membrane Associated With Proliferative Diabetic Retinopathy After Intravitreal Bevacizumab (Avastin®)
Brief Title: Intravitreal Bevacizumab for Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: koh01
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-01

CONDITIONS: Diabetic Retinopathy
Keywords: intravitreal bevacizumab; proliferative diabetic retinopathy; VEGF; PEDF
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Bevacizumab

INTERVENTIONS:
Drug: bevacizumab

SUMMARY:
Recently, intravitreal bevacizumab (Avastin) injection has gained popularity as a potential treatment of intraocular neovascularization (CNV) associated with age related macular degeneration and diabetic retinopathy. The efficacy of the drug is thought to be related with its pharmacologic blockade of VEGF.

The purpose of this study is to determine the effect of the intravitreal bevacizumab on the fibrovascular membrane associated with proliferative diabetic retinopathy by objective histologic evaluation.

The patients scheduled for vitrectomy for tractional fibrovascular membrane due to proliferative diabetic retinopathy will be randomized into two treatment groups. The one will receive conventional vitrectomy and the other group will receive intravitreal bevacizumab injection one week before the scheduled vitrectomy. The fibrovascular membrane will be excised during surgery and fixated for histologic examinations. The expression of VEGF and PEDF, a potent inhibitor of angiogenesis, will be evaluated in the fibrovascular membrane by immunohistochemistry. The results will be compared between two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Tractional retinal detachment recently involving the macula with fibrovascular membrane due to proliferative diabetic retinopathy
* Severe fibrovascular proliferation progressing after appropriate panretinal photocoagulation

Exclusion Criteria:

* Uncontrolled systemic hypertension
* Recent history of myocardiac infarction within 6 months
* Recent history of cerebrovascular accident within 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2006-12; Study Completion 2007-03

PRIMARY OUTCOMES:
expression level of VEFG
PEDG
Factor VIII

SECONDARY OUTCOMES:
complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jun Koh, Principal Investigator — Department of Ophthalmology, Yonsei University College of Medicine
Locations (1):
- Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Chen E, Park CH. Use of intravitreal bevacizumab as a preoperative adjunct for tractional retinal detachment repair in severe proliferative diabetic retinopathy. Retina. 2006 Jul-Aug;26(6):699-700. doi: 10.1097/01.iae.0000225351.87205.69. No abstract available. PMID 16829817
- [Background] Mason JO 3rd, Nixon PA, White MF. Intravitreal injection of bevacizumab (Avastin) as adjunctive treatment of proliferative diabetic retinopathy. Am J Ophthalmol. 2006 Oct;142(4):685-8. doi: 10.1016/j.ajo.2006.04.058. PMID 17011869
- [Background] Matsuoka M, Ogata N, Minamino K, Matsumura M. Expression of pigment epithelium-derived factor and vascular endothelial growth factor in fibrovascular membranes from patients with proliferative diabetic retinopathy. Jpn J Ophthalmol. 2006 Mar-Apr;50(2):116-20. doi: 10.1007/s10384-005-0294-9. PMID 16604386
- [Background] Avery RL, Pearlman J, Pieramici DJ, Rabena MD, Castellarin AA, Nasir MA, Giust MJ, Wendel R, Patel A. Intravitreal bevacizumab (Avastin) in the treatment of proliferative diabetic retinopathy. Ophthalmology. 2006 Oct;113(10):1695.e1-15. doi: 10.1016/j.ophtha.2006.05.064. PMID 17011951
- [Background] Oshima Y, Sakaguchi H, Gomi F, Tano Y. Regression of iris neovascularization after intravitreal injection of bevacizumab in patients with proliferative diabetic retinopathy. Am J Ophthalmol. 2006 Jul;142(1):155-8. doi: 10.1016/j.ajo.2006.02.015. PMID 16815267
- [Background] Bakri SJ, Donaldson MJ, Link TP. Rapid regression of disc neovascularization in a patient with proliferative diabetic retinopathy following adjunctive intravitreal bevacizumab. Eye (Lond). 2006 Dec;20(12):1474-5. doi: 10.1038/sj.eye.6702364. Epub 2006 May 5. No abstract available. PMID 16680105
- [Background] Spaide RF, Fisher YL. Intravitreal bevacizumab (Avastin) treatment of proliferative diabetic retinopathy complicated by vitreous hemorrhage. Retina. 2006 Mar;26(3):275-8. doi: 10.1097/00006982-200603000-00004. PMID 16508426